CLINICAL TRIAL: NCT03231137
Title: Socket Augmentation Using Different Platelet Concentrates, Atorvastatin Gel or Combination (Clinical and Histomorphometric Study)
Brief Title: Socket Augmentation Using Platelet Concentrates, Atorvastatin Gel or Combination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ola Mohamed Ezzatt, Lecturer Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASU-OMP-2012-9
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Alveolar Socket Preservations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- PRGF/ATV (Experimental): Included 10 patients undergoing single tooth extraction and platelet rich in growth factors fibrin scaffold loaded with Atorvastatin powder (PRGF/ATV) were placed to fill the extraction socket.
  Interventions: Combination Product: PRGF/ATV
- ATV gel (Experimental): Included 10 patients undergoing single tooth extraction and Atorvastatin gel were placed to fill the extraction socket.
  Interventions: Drug: ATV gel
- PRF (Experimental): Included 10 patients undergoing single tooth extraction and platelet rich fibrin (PRF) were placed to fill the extraction socket.
  Interventions: Biological: PRF
- PRGF (Experimental): Included 10 patients undergoing single tooth extraction and plasma rich in growth factors (PRGF) were placed to fill the extraction socket.
  Interventions: Biological: PRGF
- Control (No Intervention): Spontaneously healed socket

INTERVENTIONS:
Combination Product: PRGF/ATV — Atorvastatin (ATV) loaded on plasma rich in growth factor (PRGF) Derived Fibrin Scaffold
  Arms: PRGF/ATV
Drug: ATV gel — Atorvastatin gel
  Arms: ATV gel
Biological: PRF — Platelet rich fibrin
  Arms: PRF
Biological: PRGF — plasma rich in growth factor
  Arms: PRGF

SUMMARY:
This study was conducted to compare post-extraction augmented sockets using Atorvastatin loaded in Plasma rich in growth factors derived fibrin scaffold (PRGF/ATV) or direct application of Atorvastatin (ATV) gel or platelet rich fibrin (PRF) or (PRGF) and spontaneously healed socket (Control) both clinically and by histomorphometric analysis of formed bone quality.

DETAILED DESCRIPTION:
Ridge preservation therapies have been proposed with the aim of maintaining the hard and soft tissue dimensions of the alveolar ridge that are partially lost after tooth extraction as part of the natural physiological healing process. There are many techniques in the literature used for socket preservation as bone grafts, barrier membranes, immediate implant and socket shield. Many other techniques also are used such as bone and tissue healing promoting molecules like recombinant human bone morphogenetic protein-2 (rhBMP-2). However Autologous blood preparations like platelet-rich fibrin (PRF), and platelet rich in growth factors (PRGF) have been also introduced for socket preservation. Moreover, Statins the widely used group of cholesterol lowering drugs which also increase normal bone formation by promoting osteoblast proliferation and differentiation and protecting the from apoptosis. In addition, they reduce osteoclastogenesis by inhibiting osteoclastic differentiation. Statins increase BMP-2 gene expression and subsequently promote bone formation. in the emerging area of growth factors, there is no high-quality evidence to either support or refuse their use.

This study hypothesized that use of PRGF fibrin scaffold in socket preservation owing to its biocompatibility, ease of use, stimulation of production of growth factors and its effect on the already differentiated osteoblasts, when combined with statin with its effect on progenitor stem-cells could stimulate the differentiation of stem cells to osteoblasts, prevent bone resorption and stimulate bone formation at the extraction socket.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both genders, aged from 20 to 50 years
* 2. Patients free from any systemic diseases
* 3. Hopeless teeth indicated for extraction (badly decayed tooth, tooth contraindicated for crown preparation such as tooth with subgingival caries, broken roots, periodontally affected teeth, remaining roots) in the premolar and first molar area.
* 4. Socket type I: The facial soft tissue and buccal plate of bone are at normal levels in relation to cement-enamel junction of the pre-extracted tooth and remain intact postextraction as determined by clinical examination and periapical radiographs
* 5. Patient agreed to sign a written consent after explanation of study nature.

Exclusion Criteria:

* 1. Smokers.
* 2. Pregnant and breast feeding females.
* 3. Previous radiation, chemotherapy, or immunosuppressive treatments.
* 4. Known hypersensitivity to statin drugs.
* 5. Teeth with periapical infections, type II or III sockets or with dehiscence or fenestrations
* 6. Vulnerable groups such as (Prisoners and handicapped or mentally disabled)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06-16 (Actual); Primary Completion 2017-03-12 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Relative ridge height | baseline (immediately after extraction) - After 2 months
  (Measured from stent reference point to the crest of the buccal or palatal plate of bone)
Ridge width | baseline (immediately after extraction) - After 2 months
  (Measured from the buccal to palatal plate of bone using bone caliper)

SECONDARY OUTCOMES:
Collagen surface area | after 2 months
Average tabecular size | after 2 months

IPD SHARING:
Plan to Share IPD: Undecided